CLINICAL TRIAL: NCT04457505
Title: Risk Factors, Personalized Prognoses and 1-year Follow-ups of Patients Admitted to Spanish Intensive Care Units Due to COVID-19
Brief Title: One Year Follow-ups of Patients Admitted to Spanish Intensive Care Units Due to COVID-19
Status: Completed | Type: Observational
Sponsor: Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government)
Collaborators: Barcelona Supercomputing Center (Unknown); Carlos III Health Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: CIBERESUCICOVID
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Acute Respiratory Distress Syndrome; Severe Pneumonia; Respiratory Failure
MeSH Terms: conditions — Respiratory Distress Syndrome; Pneumonia; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — For the epigenetic study, blood samples will be gathered from 1000 patients within 48 hours after admission to the ICU. The collection and preparation of plasma samples will be done in accordance with Early Detection Research Network (EDRN) Standard Operating Procedures (National Cancer Institute, USA).
  For the study of prognostic biomarkers, concentration of biomarkers in plasma that are key to potentially useful drugs' mechanism of action in this disease will be assessed. Plasma samples will be collected from 1000 patients within 48 hours after admission to the ICU.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The latest epidemiological data published from Chine reports that up to 30% of hospital-admitted patients required admission to intensive care units (ICU). The cause for ICU admission for most patients is very severe respiratory failure; 80% of the patients present with severe acute respiratory distress syndrome (SARS) that requires protective mechanical ventilation.

Five percent of patients with SARS require extracorporeal circulation (ECMO) techniques. Global mortality data has been thus far reported in different individual publications from China. Without accounting for those patients still admitted to hospital, bona fide information (from a hospital in Wuhan) received by the PI of this project estimates that mortality of hospitalized patients is more than 10%. Evidently, mortality is concentrated in patients admitted to the ICU and those patients who require mechanical ventilation and present with SARS. As data in China was globally reported, risk factors and prognosis of patients with and without SARS who require mechanical ventilation are not definitively known. The efficacy of different treatments administered empirically or based on small, observation studies is also not known. With many still admitted at the time of publication, a recent study in JAMA about 1500 patients admitted to the ICU in the region of Lombardy (Italy) reported a crude mortality rate of 25%. The data published until the current date is merely observational, prospective or retrospective. Data has not been recorded by analysis performed with artificial intelligence (machine learning) in order to report much more personalized results. Furthermore, as it concerns patients admitted to the ICU who survive, respiratory and cardiovascular consequences, as well as quality of living are completely unknown.

The study further aims to investigate quality of life and different respiratory and cardiovascular outcomes at 6 months, as well as crude mortality within 1 year after discharge of patients with COVID-19 who survive following ICU admission. Lastly, with the objective to help personalize treatment in accordance with altered biological pathways in each patient, two types of studies will be performed: 1) epigenetics and 2) predictive enrichment of biomarkers in plasma.

Hypothesis

* A significant percentage of patients (20%) admitted to the hospital with COVID-19 infection is expected to require ICU admission, and need mechanical ventilation (80%) and, in a minor percentage (5%), ECMO.
* Patients who survive an acute episode during ICU hospitalization will have a yearly accumulated mortality of 40%. Those who then survive will have respiratory consequences, cardiovascular complications and poor quality of life (6 months).

DETAILED DESCRIPTION:
Objective and Purpose of Study

1. The main objective is to determine risks factors and prognosis of patients with COVID-19 infection who have been admitted to Spanish ICUs between the beginning and end of the pandemic in Spain. Special attention will be placed on identifying differential expression of prognostic factors based on sex.
2. The second objective is to perform a follow-up of patients within 6 months after discharge from ICU and hospital in order to determine mortality (including at 1-year mark), functional respiratory and cardiovascular consequences, and quality of life.
3. The third objective is to perform an epigenetic study in cases, in which a blood sample can be drawn. The aim of such undertaking is to define molecular signatures in liquid biopsies that can provide information regarding prognosis, and treatment monitoring and response to therapy.
4. Lastly, predictive ability of response to therapy and mortality will be assessed from a panel of protein biomarkers that participate in key physiological pathways of the disease's pathogenesis. This could, in turn, help select prospective treatments with greater potential of being successful in each patient.

Principal and Secondary Variables

1. Prior epidemiological data of the patient
2. Biological and clinical data, including treatment administered upon hospital admission
3. Biological and clinical data, including treatments administered upon and during ICU admission until either discharge from ICU or hospital, or death
4. Specific data regarding artificial ventilation and ECMO since the beginning, as well as sequentially, from intubation to either extubation or death
5. Biological and clinical data upon hospital discharge
6. Clinical follow-up of patients who survive within 6 months, including: functional respiratory tests, echocardiograms and surveys regarding quality of life
7. Intrahospital and intra-ICU mortality will be registered at 28- and 90-day marks, as well as within 6 months and 1 year
8. 1000 blood samples will be drawn for the epigenetic study The molecular profile of a non-coding RNA (ncRNA), specifically the microRNA (miRNA) pattern in liquid biopsy, will be analyzed. A circulating miRNA signature is closer to the phenotype than genomic markers and can provide information regarding epigenetic regulation, cell activation, tissue repair, and metabolic processes in addition to that afforded by clinical predictors and classic risk factors. miRNAs offer appropriate biochemical properties that are highly stable; have a long half-life in biological samples used in clinical laboratories (serum/plasma); can be efficiently and relatively rapidly quantified with high sensitivity and specificity by RT-qPCR; and can serve as a profitable tool for the assessment of risks and disease control.

All of these characteristics have led distinct authors to propose the clinical application of miRNA in either the short or medium term.

The experimental design comprises two phases. In the first approximation, a screening of non-coding RNA (ncRNA) will be performed in a sub-population of patients (n=200). The number of samples surpasses the quantity recommended for this type of studies. (Schurch y cols., RNA, 2016). A quotation will be requested for the screening of ncRNA by HTG EdgeSeq miRNA Whole Transcriptome Assay system (HTG). Using next generation sequencing (NGS), this method allows for the quantification of 2083 human candidates. All of the procedure steps will be completed in suitable physical locations in accordance with code OP No. 0028. All of the samples will be prepared in accordance with code No. 0036.

Screening results will be validated in the validation cohort (n=800) with RT-qPCR, a gold-standard technique. The budget includes material necessary for RNA extraction (miRNeasy Serum/Plasma isolation kits, Qiagen; spike-in; carrier RNA; consumables) and expression quantification of ncRNA in biofluids (RT-qPCR miRCURY LNA Universal RT microRNA PCR System kits, Qiagen; endogenous controls; consumables. Studies will be carried out at the TRRM Group facilities in the IRBLleida. The laboratory has the necessary team and material to isolate and quantify RNA, and store reagents and samples (cold stores, freezers of 20ºC and -80ºC).

9.- For the study of prognostic biomarkers, concentration of biomarkers in plasma that are key to potentially useful drugs' mechanism of action in this disease will be assessed. This quantification could provide guidance on drug usage (lymphocyte count will be obtained from a blood count):

ELIGIBILITY:
Inclusion Criteria:

* 1. Laboratory-confirmed COVID-19 infection with either real-time PCR or Next Generation Sequencing (NGS)
* 2. Admission to intensive care unit

Exclusion Criteria:

* 1. Patients admitted to COVID-19-negative ICU

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to Spanish ICUs.
Sampling Method: Probability Sample
Enrollment: 8500 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
One year mortality | At 12 months of ICU admission
  People who died after one year of follow up
Six month mortality | At 6 month of ICU admission
  People who died after one year of follow up

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Torres, PhD, Principal Investigator — Spanish Research Center for Respiratory Diseases
Locations (31):
- Spain (31):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital de Mataró, Mataró, Barcelona
  - Hospital General de Cataluña, Sant Cugat del Vallès, Barcelona
  - Hospital Infanta Margarita de Cabra, Cabra, Córdoba
  - Hospital Universitario Lucus Augusti, Lugo, Galicia
  - Hospital Son Llatzer, Palma de Mallorca, Mallorca
  - Hospital Álvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Verge de la Cinta, Tortosa, Tarragona
  - Hospital Universitario Sant Joan d'Alacant, Alicante
  - Clínica Sagrada Família, Barcelona
  - Hospital Sagrat Cor, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Vall d'Hebron University Hospital, Barcelona, Barcelona
  - Hospital Clinic, Barcelona
  - Hospital Burgos, Burgos
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital de León, León
  - Hospital Arnau de Vilanova Lleida, Lleida
  - Hospital Infanta Leonor de Madrid, Madrid
  - Hospital Universitario La Paz, Madrid
  - Complexo Hospitalario Universitario de Ourense, Ourense
  - Complejo Asistencial Universitario de Palencia, Palencia
  - Hospital Montecelo, Pontevedra
  - Hospital Universitario Salamanca, Salamanca
  - Hospital Universitari Virgen de Valme, Seville
  - Hospital Universitari de Tarragona Joan XXIII, Tarragona
  - Hospital Clínic Universitari de València, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia
  - Hospital Universitario Valladolid, Valladolid
  - Hospital Nuestra Señora de Gracia, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
All IPD anonymized that underlie results in a publication will be available after publication.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After publication
Access Criteria: Data will be available after reasoning requested.

REFERENCES:
- [Derived] Wendel-Garcia PD, Ceccato A, Motos A, Franch-Llasat D, Perez-Moreno MO, Domenech-Spanedda MF, Chamarro-Marti E, Ferrer R, Fernandez-Barat L, Riera J, Alvarez-Napagao S, Penuelas O, Lorente JA, Almansa R, Gabarrus A, de Gonzalo-Calvo D, Gonzalez J, Anon JM, Barbera C, Barberan J, Blandino-Ortiz A, Bustamante-Munguira E, Caballero J, Carbajales-Perez C, Carbonell N, Catalan-Gonzalez M, Barral-Segade P, Manez R, de la Torre MC, Diaz E, Estella A, Gallego E, Garcia-Garmendia JL, Garnacho-Montero J, Amaya-Villar R, Gomez JM, Huerta A, Jorge-Garcia RN, Loza-Vazquez A, Marin-Corral J, Martin-Delgado MC, de la Gandara AM, Martinez-Varela IY, Lopez-Messa J, Muniz-Albaiceta G, Novo MA, Penasco Y, Pozo-Laderas JC, Ricart P, Sanchez-Miralles A, Sancho S, Socias L, Sole-Violan J, Suarez-Sipmann F, Tamayo L, Trenado J, Barbe F, Torres A, Roche-Campo F; CIBERESUCICOVID Investigators. Empirical antibiotic therapy improves outcomes in mechanically ventilated patients with COVID-19: An emulated targeted trial within a prospective, multicentre cohort study. J Infect. 2025 Feb;90(2):106411. doi: 10.1016/j.jinf.2025.106411. Epub 2025 Jan 13. PMID 39814268
- [Derived] Garcia-Hidalgo MC, Gonzalez J, Benitez ID, Carmona P, Santisteve S, Perez-Pons M, Moncusi-Moix A, Gort-Paniello C, Rodriguez-Jara F, Molinero M, Belmonte T, Torres G, Labarca G, Nova-Lamperti E, Caballero J, Bermejo-Martin JF, Ceccato A, Fernandez-Barat L, Ferrer R, Garcia-Gasulla D, Menendez R, Motos A, Penuelas O, Riera J, Torres A, Barbe F, de Gonzalo-Calvo D; CIBERESUCICOVID Project (COV20/00110, ISCIII). Identification of circulating microRNA profiles associated with pulmonary function and radiologic features in survivors of SARS-CoV-2-induced ARDS. Emerg Microbes Infect. 2022 Dec;11(1):1537-1549. doi: 10.1080/22221751.2022.2081615. PMID 35603455